CLINICAL TRIAL: NCT00947804
Title: Phase 1 - Pilot Study to Validate the Simple Acute Coronary Syndrome Score; an Acute Coronary Syndrome (ACS) Risk Stratification Tool
Brief Title: Study to Validate Simple Acute Coronary Syndrome Score
Acronym: SACS Score
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: St. Joseph's Hospital, Florida (Other)
Responsible Party: Principal Investigator, Wayne Ruppert, Principal Investigator, St. Joseph's Hospital, Florida
Other Study IDs: ACS SACS Score SJH-01
Record Dates: First submitted 2009-07-26; First posted 2009-07-28 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2012-12

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute Coronary Artery Syndrome Risk Stratification Score
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1. Patients with symptoms of ACS: Patients whom present emergently to the Cardiac Catheterization Lab with current symptoms of Acute Coronary Syndrome (ACS), whom at the time of admission to the cardiac catheterization lab are believed to be suffering from STEMI, NSTEMI, or Unstable Angina, with the possible need for emergency Percutaneous Coronary Intervention (PCI), or Coronary Artery Bypass Grafting (CABG).
- 2. Patients without symptoms of ACS: Non-emergency patients presenting to the Cardiac Catheterization Lab for elective coronary angiography, and possible PCI. These are patients whom may have experienced typical or atypical ACS symptoms intermittently, and have elected to have cardiac catheterization to rule out obstructive CAD. Patients in this group will be selected randomly, with consent obtained, prior to cardiac catheterization.

SUMMARY:
The Simple Acute Coronary Syndrome (SACS) Score was developed as a Risk Stratification Tool for Acute Coronary Syndrome (ACS). It is a tool which rates a patient's: SYMPTOMS, EKG FINDINGS, RISK FACTOR PROFILE, and CARDIAC MARKERS on a scale of zero to six.

The purpose of this study is to validate the SACS Scoring tool by establishing a correlation between the score's numerical values and the degree of obstructive cardiovascular disease visualized during cardiac catheterization.

DETAILED DESCRIPTION:
Depending on whose published research is referenced, an estimated 68,000 to 136,000 people with ACS are misdiagnosed and discharged annually from our nation's emergency departments. The emotional loss to grieving family members is incalculable. The negative financial impact to families who lose their primary income providers and losses incurred by health care providers in legal expenses is also significant. Misdiagnosis of ACS is due, in part, to:

* Patients presenting with ATYPICAL symptoms of ACS
* Problems with SENSITIVITY and SPECIFICITY with the 12 Lead EKG
* Inconsistent integration of Patients' Coronary Artery Disease (CAD) Risk Factor Profile into the clinical decision making process.

One solution to improving ACS diagnostic accuracy is for clinicians to utilize an ACS Risk Stratification Tool that is proven to be highly sensitive and specific with respect to identifying patients with significant underlying CAD.

While screening approximately 50 patient case studies for inclusion in a 12 Lead EKG education curriculum, multiple incidents were noted where the patient's Modified TIMI ACS Risk Score did not accurately correlate with the patient's degree of cardiovascular disease. In several cases, the disparity between the Modified TIMI Risk Score and the patient's disease status was so great that if clinicians had considered this score in the clinical decision making process, patients would have been discharged with "clean bills of health," while actually having severe underlying CAD; scenarios that would have "set the stage" for adverse outcomes.

In the search for a more reliable ACS Risk Stratification Tool, none were found that were deemed consistently reliable enough for use as an adjunct to clinical decision making. This could be due, in part, to the fact that the tools currently available (TIMI, GRACE, PURSUIT), were primarily designed as prognostic indicators of mortality in patients diagnosed with ST Segment Elevation Myocardial Infarction (STEMI) in pharmaceutical studies - not as tools to assess the probability that ACS exists in patients presenting to the Emergency Department. This prompted the development of the SACS Score.

In approximately 50 cases informally studied to date, the SACS scoring tool produced scores that are more consistent and more predictive of the presence of obstructive CAD than the Modified TIMI Risk Score.

Our formal study will consist of at least 200 patients, which will include two groups.

GROUP 1 will consist of all Acute Myocardial Infarction (AMI) patients (STEMI / NSTEMI) treated at St. Joseph's Hospital, beginning in January, 2009 and continuing until our target number of 200 patients is obtained. In order to not delay urgent cardiac catheterization and treatment, these patients will be studied retrospectively (post cardiac catheterization and intervention).

GROUP 2 will consist of randomly selected patients whom are clinically stable at the time of cardiac catheterization. These patients will be studied prospectively. To maintain integrity of the study, these patients will be selected, with written consent obtained, prior to cardiac catheterization.

Data to be collected in all case studies (both groups) will include demographics and specific information about the patient's SYMPTOMS, EKG FINDINGS, RISK FACTOR PROFILE and CARDIAC LABS.

NOTE: ADDED JULY, 2010: To assure accuracy with respect to comparison of the SACS score to other ACS Risk Stratification scoring tools, we will only include patients in our study whose medical records reflect accurate risk factor history assessments which are consistent with TIMI risk factor assessment guidelines. For example, if it is recorded that the patient has "Family History Positive for Coronary Artery Disease," but it does not state specifically WHICH family member(s), and/or does not state the SPECIFIC CARDIAC DIAGNOSIS (such as "Acute Myocardial Infarction"), and/or does not include the AGE of the family member at the time of diagnosis, we WILL NOT include the patient in our study. A complete list of TIMI Risk Factor Assessment Guidelines TIMI guidelines can be found at www.TIMI.org,

POST CARDIAC CATHETERIZATION data will be classified into categories based on cath lab findings:

1. No visible CAD present
2. Mild-to-moderate plaquing without obstructive CAD. No catheter-based or surgical intervention was performed. Number of lesions, location(s), and percentage(s) of arterial obstruction will be specified.
3. Significant obstructive CAD present. Number of lesions, location(s), and percentage(s) of arterial obstruction and intervention(s) performed will be specified.
4. Acute total occlusion of coronary artery requiring emergency intervention. Location of lesion and intervention(s) performed will be specified.

Regression Analysis of 126 data points collected from each patient will be used to establish relationships between score values and the degree of obstructive CAD present.

We believe that once scientifically validated, the SACS Score will become a useful tool to aid medical professionals in reducing the incidence of patients whom are misdiagnosed with respect to ACS.

ELIGIBILITY:
Inclusion Criteria:

* Must be mentally competent with ability to articulate symptoms and risk factor profile

Exclusion Criteria:

* Renal disease
* When unable to obtain all required data sets (SYMPTOMS, EKG, TIMI RISK FACTOR PROFILES, CARDIAC LABS)
* EKG displays DELTA WAVES consistent with Wolff-Parkinson-White Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients presenting to the cardiac catherization suite whom have experienced ACS symptoms within the past thirty days.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-08; Primary Completion 2013-12 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
PRESENCE or ABSENCE of obstructive CAD as discovered during non-investigative coronary angiography in the Cardiac Catheterization Lab. | Within 24 hours of: a) arrival in Emergency Department, or b) admission to the hospital

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Ruppert, CVT, Principal Investigator — St. Joseph's Hospital, Tampa, FL; Humberto Coto, MD, FACC, Study Director — St. Joseph's Hostpial, Tampa, Florida; Xavier E Prida, MD, FACC, Study Director — St. Joseph's Hospital, Tampa, Florida; Charles Sand, MD, FACEP, Study Director — St. Joesph's Hospital, Tampa, FL
Locations (1):
- St. Joseph's Hospital, Tampa, Florida, United States